CLINICAL TRIAL: NCT03878212
Title: Effects of mHealth on Promoting Self-care Health Management Among Older Adults in the Community: A 3-arm Randomized Controlled Trial
Brief Title: Effects of mHealth on Promoting Self-care Health Management Among Older Adults in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Principal investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: mHSC-01
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Telemedicine
Keywords: mHealth; app
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mHealth+I (Experimental): This group of participants will receive a proactive mHealth with interactivity program which includes two main elements: 1) mHealth application designed by the research team with the information technological support by Smartone and 2) nurse case management supported by a social service team
  Interventions: Other: mHealth application with interactivity
- mHealth (Active Comparator): The mHealth group will have access to the health content on the mHealth platform. This group 2018 HMRF Open Call Proposal Section 13: Proposed Research Project 5 will enjoy the same content and client-initiated help if needed. Same as the above group, the client is invited to use the mHealth application. A reminder message will pop up on the screen of smartphone when participants have not used it for more than one week. The participants are encouraged to read the self-care information that is featured in the app. There is a button for the client-imitated call if they would like to consult a nurse.
  Interventions: Other: mHealth application
- Control (No Intervention): All groups will receive usual community services. The study district provides community-based health talks and basic health checks such as measuring blood pressure and blood glucose that are accessible to all residents, and their participation is voluntary. Both health and social services are available in the community for those who need help, including referral for further help if appropriate. These services are however episodic with design for continuity of care. No mHealth application will be provided to the participants in this group but the individuals are free to do their own surfing for e-health information.

INTERVENTIONS:
Other: mHealth application with interactivity — a mHealth device with interactivity with nurse case manager
  Arms: mHealth+I
Other: mHealth application — a mHealth device
  Arms: mHealth

SUMMARY:
Many of the existing mobile health (mHealth) apps designed in a reactive care approach, in which people do not receive individualized care until they consulted health care professionals through the apps. This proposal endeavors to develop a proactive mHealth application on promoting self-care ability and health among older adults to examine the differential benefits of adding nurse interaction supported by an integrated health-social partnership model in the use of mHealth.

DETAILED DESCRIPTION:
Objectives: Many of the existing mobile health (mHealth) apps designed in a reactive care approach, in which people do not receive individualized care until they consulted health care professionals through the apps. This proposal endeavors to develop a proactive mHealth application on promoting self-care ability and health among older adults to examine the differential benefits of adding nurse interaction supported by an integrated health-social partnership model in the use of mHealth.

Hypothesis to be tested: There is no difference in self-management outcomes, individual and societal benefits between the subjects receiving mHealth+Interactivity, mHealth, and usual care.

Design and subjects: This is a single-blinded, three-armed randomized controlled trial. The subjects are people who are aged 60 or above with chief complaints of either pain, hypertension, or diabetes mellitus.

Instruments: mHealth application designed by the research team with the information technological support by Smartone.

Interventions: mHealth with interactivity group receives both mHealth app and nurse case management supported by a social service team in community. mHealth group will have access to health content on mHealth platform only. Usual care group receives usual community services.

Main outcome measures: Self-management outcomes (self-efficacy, pain score, blood pressure, capillary blood glucose), individual (quality of life, depression) and societal benefits (institutionalization and health service utilization).

Data analysis: Generalized Estimating Equation (GEE) is used to determine the between-group effects, within-group effects, and the interaction effects.

Expected results: Older adults would benefit from supported self-care equipping them with sufficient knowledge, skills and confidence to lead to relatively independent life at home.

ELIGIBILITY:
Inclusion Criteria:

* people who are aged 60 or above
* with chief complaints of either pain, hypertension, or diabetes mellitus
* living within the service areas and (4) using smartphone

Exclusion Criteria:

* already engaged in other mHealth programs
* diagnosed with psychiatric problems
* bed-bound
* living in area with no internet coverage

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Quality of life (general well-being of individual) | 3-month
  Quality of life will be measured by SF-12v2 (physical and psychological component) version which has been translated, validated and proven reliable for use among the Hong Kong Chinese population.This questionnaire is a generic measure, as opposed to one that targets a specific age and disease. It has shown useful in Chinese elderly patients. The scale ranged from 0 to 100, with 50 indicating the standardized norm scale

SECONDARY OUTCOMES:
depression | 3-month
  Depression will be measured by the Chinese version of the Geriatric Depression Scale. Good validity and reliability were reported in this scale, with criterion-related validity 0.95 and test-retest reliability 0.85 among the elderly Chinese population. The questionnaire consists of 15 questions which are used to explore the feelings of participants with the dichotomous answers. The scale has ranged from 0 to 15, higher scores indicated higher depressive severity.
self-efficacy | 3-month
  Self-efficacy will be measured by General Self-Efficacy Scale. This scale is used to determine how people judge their ability to handle difficult situations or solve their own problems, and thus can be a way to assess the effectiveness of empowerment programs. All 10-item in the Chinese version are rated on a 4-point Likert scale ranging from 1= not at all true to 4= exactly true. Scores on the scale are summated and higher scores indicate greater self-efficacy.Measuring general self-efficacy can provide a way to evaluate the effectiveness of empowerment interventions.
pain score | 3-month
  Pain score is measured by Visual Analog Scale that installed in the app. Pain score is ranging from 0 (no pain) to 10 (severe pain).
blood pressure | 3-month
  Blood pressure measurement will be performed after 10 minutes of sitting rest. A standard electronic sphygmomanometer will be used to measure supine blood pressure on the right arm of each candidate (unless contraindicated).
capillary blood glucose | 3-month
  Capillary blood glucose level will be measured by a standard capillary glucose meter.
health service utilization | 3-month
  Health service utilization will be measured by the number of attendance to government out-patient clinics (GOPC), and number of unscheduled visits to the emergency department and hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, Master, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Lutheran Group of social service, Hong Kong, Siu Sai Wan, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AKC, Bayuo J, Wong FKY, Chow KKS, Wong SM, Lau ACK. The Synergistic Effect of Nurse Proactive Phone Calls With an mHealth App Program on Sustaining App Usage: 3-Arm Randomized Controlled Trial. J Med Internet Res. 2023 May 1;25:e43678. doi: 10.2196/43678. PMID 37126378
- [Derived] Wong AKC, Wong FKY, Chow KKS, Wong SM, Bayuo J, Ho AKY. Effect of a Mobile Health Application With Nurse Support on Quality of Life Among Community-Dwelling Older Adults in Hong Kong: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2241137. doi: 10.1001/jamanetworkopen.2022.41137. PMID 36350651
- [Derived] Wong AKC, Wong FKY, Bayuo J, Chow KKS, Wong SM, Lee AYL. A randomized controlled trial of an mHealth application with nursing interaction to promote quality of life among community-dwelling older adults. Front Psychiatry. 2022 Oct 18;13:978416. doi: 10.3389/fpsyt.2022.978416. eCollection 2022. PMID 36329920